CLINICAL TRIAL: NCT05181605
Title: Survival Analysis After Neoadjuvant Therapy in Patients With Resectable Pancreatic Cancer and Risk Factors
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de investigación e innovación biomédica de Cádiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICI20-00047
Record Dates: First submitted 2021-11-08; First posted 2022-01-06 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2021-11

CONDITIONS: Pancreatic Adenocarcinoma; Pancreatic Cancer Resectable
MeSH Terms: interventions — folfirinox; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: No intervention - standard of care (No Intervention): A group of patients with pancreatic carcinoma plus risk factors will be treated per standard of care on site (surgical resection and adjuvant therapy)
- Experimental: Neoadyuvant therapy plus standard of care (Experimental): A group of patients with pancreatic carcinoma plus risk factors will be treated with neoadjuvant therapy before surgical resection and adjuvant therapy
  Interventions: Drug: Folfirinox and Stereotactic Body Radiotherapy

INTERVENTIONS:
Drug: Folfirinox and Stereotactic Body Radiotherapy — Neoadjuvant treatment is composed of folfirinox plus stereotactic body radiotherapy
  Arms: Experimental: Neoadyuvant therapy plus standard of care

SUMMARY:
Resectable Pancreatic Cancer represents an important health problem not because of its incidence, but because of its high mortality. Diagnosis in the initial stages is difficult, since the first symptoms of disease are often nonspecific. Only 15 - 25% of patients would undergo surgery with curative resection at the time of initial diagnosis. There is no an effective screening test for early diagnosis. A characteristic that defines the pancreatic adenocarcinoma is its aggressiveness. There is a high prevalence of patients who present metastatic disease at the time of diagnosis, therefore, it is evident that this tumor is capable of early systemic spread. Starting from the high prevalence of patients who experience metastatic disease shortly after undergoing a potentially curative resection, it is likely that at the time of diagnosis, the majority of pancreatic adenocarcinomas have progressed to systemic spread. The overall 5-year survival of the patients is 5.8% and has not increased in the last 10 years; the 5-year survival rate after curative surgery is not higher (7%). Patients with resectable adenocarcinoma of the pancreas, only 15% are diagnosed at an early stage (T1, T2 without lymph node involvement), these are associated with improved survival. The surgery required to treat pancreatic cancer is aggressive. To optimize results, you need to follow a series of guidelines strictly. The current standard treatment regimen for resectable pancreatic adenocarcinoma is based on surgery plus adjuvant chemotherapy. With all this, the survival rate at five years after surgery is not greater than 7%, and in addition, there is a high percentage of patients who experience metastatic disease after surgical resection with curative intent. This indicates that at the time of diagnosis, it is likely that most adenocarcinomas pancreatic diseases have progressed to systemic spread. For this reason, for years there is a growing interest in investigating new therapeutic approaches, such as the role of neoadjuvant therapy.

DETAILED DESCRIPTION:
Disease: Pancreatic cancer resectable plus risk factors

Hypothesis: The overall survival in patients treated with neoadjuvant chemotherapy before surgery -resection- plus adjuvant chemotherapy is higher than in patients treated per standard of care (only with adjuvant chemotherapy after surgery)

Objectives:

Main objective: To assess overall survival in patients treated with neoadjuvant chemotherapy before surgery-resection and adjuvant chemotherapy vs patients treated only with adjuvant chemotherapy after surgery-

Secondary objectives: To assess in both patients (experimental vs control arms): - Progression free survival - Number of completed cycles fo chemotherapy - Local and metastatic recurrence - Post-surgical morbidity - Resection rate R0 - Safety of the neoadjuvant chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients diagnosed with resectable pancreatic adenocarcinoma plus risk factors
* 2. Histological diagnosis of pancreatic adenocarcinoma by fine needle aspiration (FNA) performed by Echoendoscopy.
* 3. Patients who have not received prior therapy for pancreatic cancer.
* 4. Biliary drainage prior to neoadjuvant treatment.
* 5. Age> 18 years and <70 years.
* 6. No history of cerebrovascular accident (CVA) or myocardial infarction (MI) in 6 months prior to neoadjuvant treatment.
* 7. Women of childbearing potential and sexually active men must agree to the use of appropriate contraceptive methods (hormonal, barrier, or abstinence) prior to study enrollment and during study participation.
* 8. Patients should have normal organs and spinal function.
* 9. Ability to understand, and willingness to sign a written informed consent document

Exclusion Criteria:

* 1. Patients with resectable pancreatic adenocarcinoma without risk factors.
* 2. Patients with borderline pancreatic adenocarcinoma.
* 3. Patients with locally advanced pancreatic adenocarcinoma.
* 4. Patients with metastatic adenocarcinoma of the pancreas.
* 5. Patients who have received prior chemotherapy or radiotherapy for pancreatic adenocarcinoma
* 6. Pathological subtypes other than adenocarcinoma.
* 7. Patients included in a clinical trial in a period of 6 months prior to inclusion in this study.
* 8. A past history of allergic reaction attributed to 5-FU, leucovorin, Irinotecan or Oxaliplatin or to compounds of similar chemical or biological composition.
* 9. Uncontrolled breakthrough disease.
* 10. Patients with HIV, HBV and HCV positive and currently under antiretroviral therapy.
* 11. Other active malignancies
* 12. Pre-existing neuropathy, grade > 1.
* 13. Inflammatory bowel disease that is not controlled, or under current active therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-04-15 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | through study completion, an average of 3 year
  Weeks until death

SECONDARY OUTCOMES:
Period until recurrence disease | through study completion, an average of 3 year
  Weeks until progression disease (local or metastatic recurrence)
Number of completed chemotherapy cycles | during chemiotherapy completion, an average of 3 year
  Number of completed chemotherapy cycles
Progression disease | through study completion, an average of 3 year
  Progression disease per RECIST 1.1
Post-surgical events (if any) | through post-surgical period (6 months)
  physiological parameter for post-surgical events (if any)
Post-surgical events (if any) | through post-surgical period (6 months)
  Number of post-surgical events (if any)
Adverse events | through study completion, including follow up period, an average of 4 years
  Type and number of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: María Jesús Castro Santiago, Study Director — Hospital Universitario Puerta del Mar
Locations (1):
- Hospital Puerta del Mar, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: Yes
The study results will be published in scientific oncologyc journal and available in PubMed and clinicaltrials websites
Supporting Information: Study Protocol
Time Frame: We hope data are available in Dec-2025 (anticipated).